CLINICAL TRIAL: NCT04166435
Title: Temozolomide and Olaparib for O6-Methylguanine DNA Methyltransferase Promoter Hypermethylated Colorectal Cancer
Brief Title: TMZ + Olaparib for MGMT Hypermethylated Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000026632
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Results first posted 2023-01-30 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Temozolomide; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Temozolomide + Olaparib (Experimental): Temozolomide (75 mg/m2 orally on days 1-7 every 3 weeks) + Olaparib (150 mg orally twice daily days 1-21) in a 21-day cycle.
  Interventions: Drug: Temozolomide + Olaparib

INTERVENTIONS:
Drug: Temozolomide + Olaparib — Temozolomide (75 mg/m2 orally on days 1-7 every 3 weeks) + Olaparib (150 mg orally twice daily days 1-21) in a 21-day cycle.

SUMMARY:
This is a Phase II, non-randomized, open-label study to evaluate temozolomide in combination with olaparib in patients with MGMT promoter hypermethylated advanced colorectal cancer.

DETAILED DESCRIPTION:
This is a Phase II, non-randomized, open-label study to evaluate temozolomide in combination with olaparib in patients with MGMT promoter hypermethylated advanced colorectal cancer. Patients will receive temozolomide orally daily on days 1-7 and olaparib twice daily continuously. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. After completion of study treatments patients are followed up at 30 days, and for patients that come off treatment for reasons other than disease progression, clinical assessments will continue every 6 weeks for the first year and every 12 weeks after the first year.

PRIMARY OBJECTIVES:

I. To determine the efficacy of TMZ in combination with olaparib in subjects with MGMT promoter hypermethylated advanced colorectal cancer by the overall response rate.

SECONDARY OBJECTIVES:

I. To determine the safety of TMZ in combination with olaparib. II. To estimate the progression free survival (PFS). III. To estimate overall survival (OS).

EXPLORATORY OBJECTIVES:

I. Characterize NGS profiling, patterns of DNA methylation, gene expression, and develop MGMT expression assays.

II. Correlate molecular features with Gamma H2AX with response. III. Establish organoids for MGMT promoter hypermethylated colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).
* Provision of signed and dated, written informed consent form prior to any mandatory study specific procedures, sampling, and analyses.
* For inclusion in i) the optional exploratory genetic research and ii) the optional biomarker research, patients must fulfill the following criteria:

  * Provision of informed consent for genetic research prior to collection of sample
  * Provision of informed consent for biomarker research prior to collection of sample **If a patient declines to participate in the optional exploratory genetic research or the optional biomarker research, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study.
* Individuals who are healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Individuals with histologically proven relapsed/refractory mismatch repair proficient / microsatellite stable metastatic colorectal adenocarcinoma.
* MGMT promoter hypermethylation on pre-screening.
* Patients must have had recurrence, progression or intolerance to standard therapy consisting of at least 2 prior standard regimens (containing a fluoropyrimidine plus a platinum analogue and/or irinotecan) for metastatic disease. In the case where all chemotherapy agents are used concurrently (I.e. FOLFOXIRI +/- Bevacizumab) 1 prior treatment regimen is acceptable after discussion with the principal investigator. Relapse within 6 months of completing adjuvant chemotherapy is considered one line of therapy in the metastatic setting.
* Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

  * Haemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5x ULN.
  * Patients must have creatinine clearance estimated of ≥51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test :
  * Estimated creatinine clearance = (140-age [years]) x weight (kg) (x F)° / serum creatinine (mg/dL) x 72

    * where F=0.85 for females and F=1 for males.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Patients must have a life expectancy ≥ 16 weeks.
* At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.

  * Postmenopausal is defined as:
  * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
  * Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50
  * radiation-induced oophorectomy with last menses >1 year ago
  * chemotherapy-induced menopause with >1 year interval since last menses
  * surgical sterilisation (bilateral oophorectomy or hysterectomy)
* Male patients must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception ([see appendix C for acceptable methods]) if they are of childbearing potential.

Exclusion Criteria:

* Other malignancy unless curatively treated with no evidence of disease for ≥5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma.
* Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
* Persistent toxicities (Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
* Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Patients with known active hepatitis (i.e. Hepatitis B or C).
* Active hepatitis B virus (HBV) is defined by a known positive HBV surface antigen (HBsAg) result. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible.
* Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Any previous treatment with PARP inhibitor, including Olaparib.
* Any previous treatment with temozolomide or other monofunctional alkylating agent.
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib and temozolomide is 2 weeks.
* Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib and temozolomide is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable, for timing refer to inclusion criteria related to "Patients must have had recurrence, progression or intolerance to standard therapy...").
* Participation in another clinical study with an investigational product administered in the last 28 days.
* Subjects with a known hypersensitivity to temozolomide, olaparib, any of the recipients of either product, or the combination.
* Patients with a known hypersensitivity to the combination/comparator agent.
* Involvement in the planning and/or conduct of the study
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
* Previous enrollment in the present study.
* Breast feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cecchini, MD, Principal Investigator — Assistant Professor of Medicine (Medical Oncology) Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Temozolomide + Olaparib
Started | 11
Completed | 9
Not Completed | 2
Not completed — 2 patients ineligible for response | 2

BASELINE CHARACTERISTICS:
Arm/Group | Temozolomide + Olaparib
Number analyzed (Participants) | 9
Age, Customized [Median (Full Range); unit: years] | 59 [45 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8
  Black | 1
Region of Enrollment [Number; unit: participants]
  United States | 9
ECOG performance status [Count of Participants; unit: Participants] — Graded according to the ECOG Performance Status Scale 0-5
  Participants
    0-Fully active, able to carry on all pre-disease performance without restriction | 3
    1-No physically strenuous activity but ambulatory and can carry out light or sedentary activities | 6
    2-Capable of selfcare but can't carry out any work activities; up to about 50% of waking hours | 0
    3-Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours | 0
    4-Completely disabled; cannot carry on any selfcare; totally confined to bed or chair | 0
    5-Dead | 0
Side of primary tumor [Count of Participants; unit: Participants] — Right side defined as tumors primary to splenic flexure
  Participants
    Left | 4
    Right | 5
Tumor Grade [Count of Participants; unit: Participants]
  Poorly differentiated | 3
  Moderately differentiated | 6
Molecular Results [Count of Participants; unit: Participants]
  KRAS mutated | 7
  KRAS/RAF wildtype | 2
Number of prior therapies [Count of Participants; unit: Participants]
  2 | 2
  ≥ 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: To determine the efficacy of TMZ in combination with olaparib in subjects with MGMT promoter hypermethylated advanced colorectal cancer. The overall response rate (ORR) was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) before and after treatment. Complete Response (CR): disappearance of all target lesions, Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD). Clinical Benefit is defined as the sum of CR, PR, or SD post treatment from the start of treatment.
Time Frame: Up to 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Temozolomide + Olaparib
Number analyzed (Participants) | 9
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 5
  Progressive Disease | 4

2. Secondary Outcome: Count of Participants With Adverse Events Greater or Equal to 3
Description: To determine the safety of TMZ in combination with olaparib, the number of participants with ≥ grade 3 treatment related adverse events by CTCAE v5.0 coding will be assessed.
Time Frame: Up to 2 years from last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Temozolomide + Olaparib
Number analyzed (Participants) | 9
Participants | 7

3. Secondary Outcome: Progression Free Survival
Description: To estimate the progression free survival (PFS), patients will be followed for up to 24 months.
Time Frame: Up to 2 years from last treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide + Olaparib
Number analyzed (Participants) | 9
months | 3 [2.1 to NA] — upper limit was not reached

4. Secondary Outcome: Overall Survival
Description: To estimate overall survival (OS), patients will be followed for up to 24 months.
Time Frame: Up to 2 years from last treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide + Olaparib
Number analyzed (Participants) | 9
months | 9.4 [6.7 to NA] — upper limit not reached

ADVERSE EVENTS:
Time Frame: up to 2 years
Arm/Group | Temozolomide + Olaparib
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide + Olaparib (N=9)
Nausea (Gastrointestinal disorders) | 1 (1) — one patient nausea/vomiting that was related to underlying disease
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Temozolomide + Olaparib (N=9)
Nausea (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
White blood cell decreased (Investigations) | 6
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 5
Anemia (Blood and lymphatic system disorders) | 4
Lymphocyte count decreased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT04166435/Prot_SAP_000.pdf